CLINICAL TRIAL: NCT04005742
Title: The Biomarkers Of RIsk of Colorectal Cancer (BORICC) Follow-Up (BFU) Study
Acronym: BFU
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 207081
Record Dates: First submitted 2019-06-25; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; biomarkers; cancer risk; cancer prevention; ageing; diet; obesity; physical activity; colorectal adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Participants recruited to the healthy arm of the BORICC Study (BORICC1) at baseline.
- Polyp: Participants recruited to the polyp arm of the BORICC Study (BORICC2) at baseline, with a prior history of polyps.

SUMMARY:
Worldwide, colorectal cancer is the 3rd most common cancer; risk increases with age and is modified by lifestyle factors notably diet, physical activity and obesity. The BORICC Follow-Up (BFU) Study is a 12+ year follow-up of participants recruited to the Biomarkers of Risk of Colon Cancer (BORICC) Study. This longitudinal study will investigate associations between ageing and lifestyle factors and a panel of molecular biomarkers linked with colorectal cancer risk.

DETAILED DESCRIPTION:
The BORICC Follow-Up (BFU) Study builds on the findings from the BORICC Study where the investigators observed associations between age and nutritional factors, including selenium and folate, and biomarkers of colorectal health.

The BFU Study will investigate the relationships between ageing (12+ years) and such biomarkers longitudinally. It is anticipated that the project will produce novel data on (i) changes in biomarkers of colorectal cancer risk with age and (ii) the effects of obesity and lifestyle factors on biomarkers of colorectal cancer risk. These biomarkers include differentially expressed proteins, DNA methylation markers and inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* Took part in the BORICC Study at baseline (recruited 2005/6)

Exclusion Criteria:

* Unable to travel to the hospital to attend study visit
* Unable to provide informed written consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who took part in the BORICC Study at baseline (2005/06) will be invited to participate in the BFU Study. This will include both participants recruited to the BORICC1 arm (healthy participants) and those recruited to the BORICC2 arm, with a prior history of polyps.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Faecal calprotectin concentrations (marker of local inflammation) | 12 years (on average)
Serum high-sensitivity C-Reactive Protein concentrations (marker of systemic inflammation) | 12 years (on average)

SECONDARY OUTCOMES:
Gut microbiota (analysed in stool samples) | 12 years (on average)
  Abundance and diversity of the gut microbiota assessed in stool samples
Faecal short-chain fatty acid concentrations | 12 years (on average)
  Concentrations and proportions of short-chain fatty acids e.g. acetate, propionate and butyrate
DNA methylation in rectal mucosal biopsies(% methylation) | 12 years (on average)
  Target gene and global methylation (LINE-1) in rectal mucosal biopsies
Target gene expression in rectal mucosal biopsies | 12 years (on average)
  Expression of genes related to inflammation and the WNT signalling pathway in rectal mucosal biopsies
microRNA expression in rectal mucosal biopsies | 12 years (on average)
  Expression of microRNAs in rectal mucosal biopsies
Colonic crypt cell proliferative state | 12 years (on average)
  Total number and distribution of proliferating cells in rectal mucosal crypts
Colonic crypt cell dimensions | 12 years (on average)
  Height (length) and width rectal mucosal crypts
Markers of mitochondrial function and structure in rectal mucosal biopsies | 12 years (on average)
  Markers of mitochondrial function and structure in rectal mucosal biopsies such as oxidative phosphorylation proteins, namely complex I and IV
Parathyroid hormone in plasma | 12 years (on average)
25-hydroxy vitamin D concentrations in serum | 12 years (on average)
Vitamin B12 concentrations in serum | 12 years (on average)
Folate concentrations in serum | 12 years (on average)
Triglycerides in plasma | 12 years (on average)
HDL cholesterol in plasma | 12 years (on average)
LDL cholesterol in plasma | 12 years (on average)
Total cholesterol in plasma | 12 years (on average)
Glucose in plasma | 12 years (on average)
HbA1c in whole blood | 12 years (on average)

OTHER OUTCOMES:
Timed-up and go test time | 12 years (on average)
Hand grip strength using dynamometer | 12 years (on average)
Heel bone density using Achilles heel ultrasound device | 12 years (on average)
Body weight in kg | 12 years (on average)
BMI in kg/m2 (calculated from height and weight) | 12 years (on average)
Height in cm | 12 years (on average)
Body fat percentage | 12 years (on average)
  Measured using Tanita Bioimpedance scales
Habitual dietary intake assessed using Food Frequency Questionnaire | 12 years (on average)
Physical activity levels assessed using Lifestyle Questionnaire | 12 years (on average)
Physical activity levels assessed using accelerometer | 12 years (on average)
Sedentary behaviour assessed using Lifestyle Questionnaire | 12 years (on average)

CONTACTS AND LOCATIONS:
Overall Officials: John Mathers, Principal Investigator — Newcastle University
Locations (1):
- North Tyneside General Hospital, North Shields, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No